CLINICAL TRIAL: NCT05541861
Title: An Exploratory Phase I, Randomized, Observer-blind, Active-controlled, Dose-escalation Trial Evaluating the Safety, Tolerability, and Immunogenicity of an Investigational RNA-based SARS-CoV-2 Vaccine in COVID-19 Vaccine Experienced Healthy Adults
Brief Title: Safety and Effects of an Investigational COVID-19 Vaccine as Booster in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: BNT162-21
Record Dates: First submitted 2022-09-14; First posted 2022-09-15 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: Ribonucleic acid (RNA) vaccine; Vaccine; Active immunization to prevent coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Dose 1 was given observer-blind for Cohorts 1 to 4 and open-label for Cohort 5. Dose 2 was given open-label for Cohorts 1 to 5.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) (Experimental): Participants aged 18-55 years received an intramuscular injection of BNT162b2 Bivalent 30 mcg along with BNT162b4 5 mcg at Day 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg; Biological: BNT162b4 5 mcg
- Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) (Experimental): Participants aged 18-55 years received an intramuscular injection of BNT162b2 Bivalent 30 mcg along with BNT162b4 10 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Bivalent 30 mcg along with BNT162b4 10 mcg again as Dose 2 at 6 to 7 months after Dose 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg; Biological: BNT162b4 10 mcg
- Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) (Experimental): Participants aged 18-55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 15 mcg at Day 1, Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 15 mcg again as Dose 2 at 6 to 7 months after Dose 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg; Biological: BNT162b4 15 mcg; Biological: BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg
- Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) (Experimental): Participants aged >55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 15 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 15 mcg again as Dose 2 at 6 to 7 months after Dose 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg; Biological: BNT162b4 15 mcg; Biological: BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg
- Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) (Experimental): Participants aged 18-55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 30 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 30 mcg again as Dose 2 at 6 to 7 months after Dose 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg; Biological: BNT162b4 30 mcg; Biological: BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg
- Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) (Experimental): Participants aged >55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 30 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 30 mcg again as Dose 2 at 6 to 7 months after Dose 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg; Biological: BNT162b4 30 mcg; Biological: BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg
- Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) (Active Comparator): Participants aged 18-55 years received one intramuscular injection of BNT162b2 30 mcg at Day 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg
- Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years) (Active Comparator): Participants aged >55 years received one intramuscular injection of BNT162b2 30 mcg at Day 1.
  Interventions: Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg
- Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) (Experimental): Participants aged 18-55 years received two intramuscular injections of BNT162b4 30 mcg at Day 1 and 2 months post-Dose 1, respectively.
  Interventions: Biological: BNT162b4 30 mcg

INTERVENTIONS:
Biological: BNT162b2 Bivalent (original/Omicron BA.4/BA.5) 30 mcg — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years); Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years); Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years); Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years); Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years); Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years); Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years); Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Biological: BNT162b4 5 mcg — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years)
Biological: BNT162b4 10 mcg — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years)
Biological: BNT162b4 15 mcg — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years); Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years)
Biological: BNT162b4 30 mcg — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years); Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years); Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Biological: BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection.
  Arms: Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years); Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years); Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years); Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years)

SUMMARY:
This was an exploratory Phase I, randomized, observer-blind, active-controlled, dose-escalation trial to evaluate four dose levels (DLs) of BNT162b4 given in combination with BNT162b2 Bivalent (original/Omicron BA.4/BA.5) to select a safe and tolerable dose and to evaluate BNT162b4 + BNT162b2 Bivalent (original/Omicron BA.4/BA.5) when given as Dose 1 and Dose 2 (booster) in Cohorts 1 and 2 and BNT162b4 + BNT162b2 Monovalent (OMI XBB.1.5) when given as Dose 2 (booster) in Cohorts 3a, 3b, 4a, and 4b, and 30 microgram (mcg) BNT162b4 when given alone as Dose 1 and Dose 2 in Cohort 5.

The trial used a staggered dosing process schema, i.e., enrollment into the next higher dose level was done sequentially and subject to safety data from the previous dose levels, with sentinel participants in Cohorts 1, 2, 3a, and 4a. Cohort 3b investigating the same dose level as cohort 3a but in participants aged >55 years was opened after safety data for participants aged 18-55 years in Cohort 3a had been reviewed. Enrollment into Cohorts 4a and 4b was opened after safety data for Cohort 3a and 3b had been reviewed. Cohort 5 participants were not randomized and received two doses of BNT162b4 alone after which a safety review was performed after all participants received Dose 2 in this cohort.

BNT162b4 plus BNT162b2 Bivalent (original/Omicron BA.4/BA.5)/Monovalent (OMI XBB.1.5) was co-administered (as a single injection).

BNT162b4 alone was administered as a single injection.

ELIGIBILITY:
Inclusion Criteria (applicable to all dose groups unless specified otherwise):

* Had given informed consent by signing and dating the informed consent form (ICF) before initiation of any trial-specific procedures.
* Were willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions, e.g., to follow good practices to reduce their chances of being infected or spreading COVID-19, and other requirements of the trial. This included that they were able to understand and follow trial-related instructions.
* Were aged 18 years and older at randomization (Cohorts 1-4) or 18 to 55 years (Cohort 5), had a body mass index over 18.5 kg/m^2 and under 35 kg/m^2 (Cohorts 1-4) and under 30 kg/m^2 (Cohort 5), and weighed at least 50 kg at Visit 0.
* Were healthy, in the clinical judgment of the investigator based on participant-reported medical history data, and physical examination, 12-lead ECG, vital signs, and clinical laboratory test outcomes at Visit 0.

  * Note: Healthy participants with pre-existing stable disease (e.g., obesity), defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 84 days before Visit 0, could be included.
* Agreed not to enroll in another trial with an IMP starting from Visit 0 and until 168 days (Cohorts 1-4) and 90 days (Cohort 5) after receiving the last IMP dose. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only): If 168 days after the participant's first IMP dose had passed before they consented to Dose 2, they should have agreed to not enroll in another trial from the time of consent to Dose 2 until 168 days after receiving Dose 2 of the IMP.
* Agreed not to be vaccinated with:

  * Non-trial vaccines (except COVID-19 vaccines, as per next sub-bullet) starting 28 days prior to the Dose 1 and until 28 days after receiving of the last IMP dose. Seasonal influenza vaccine is allowed; however, it should be given at least 14 days before or after any administration of IMP. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only): If 28 days after the participant's first IMP dose had passed before they consented to continue Dose 2, they should not have been vaccinated with non-trial vaccines starting from the time of consent to Dose 2 and until 168 days after receiving the Dose 2 of the IMP.
  * Non-trial COVID-19 vaccines starting at least 90 days prior to the Visit 1 and until completion of the participant's last trial visit (Cohorts 1-4) and until 28 days post-Dose 2 (Cohort 5 only).
* Had been vaccinated with at least three doses of an RNA-based COVID-19 vaccine authorized in the United States (US) before Visit 0. The last COVID-19 RNA vaccine dose must have been administered at least 90 days before Visit 1.

  * Note: Documented confirmation of prior COVID-19 vaccine receipt must be obtained prior to randomization (Cohorts 1-4) or prior to Visit 1 (Cohort 5 only).
* Had negative human immunodeficiency virus (HIV) -1 and HIV-2 test results at Visit 0.
* Had negative Hepatitis B surface antigen test results at Visit 0.
* Had negative anti-Hepatitis C virus (HCV) antibodies, or negative HCV polymerase chain reaction test results if the anti-HCV was positive at Visit 0.
* Participants of childbearing potential (POCBP) that had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test result at Visit 0 and negative urine pregnancy test results prior to receiving Dose 1, additionally for Cohort 5 only, a negative urine pregnancy test result prior to receiving Dose 2. Participants born female that were postmenopausal or permanently sterilized (verified by medical records) were not considered POCBP. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only): POCBP that had a negative urine pregnancy test results prior to receiving Dose 2.
* POCBP who agreed to practice a highly effective form of contraception and required their male sexual partners to use condoms with a spermicidal agent, starting at Visit 0 and continuously until 28 days after receiving the last IMP dose. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only) : If 28 days after the participant's first IMP dose had passed before they consent to continue Dose 2, they should have a negative urine β-HCG pregnancy test result at Visit 7 and agree to practice a highly effective form of contraception and required their male sexual partners to use condoms with a spermicidal agent, starting from the time they consent to Dose 2 and continuously until 28 days after receiving Dose 2 of IMP.
* POCBP who agreed not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting at Visit 0 and continuously until 28 days after receiving the last IMP dose. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only): If 28 days after the participant's first IMP dose had passed before they consented to continue Dose 2, they should have agreed not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting from the time they consented to Dose 2 and continuously until 28 days after receiving Dose 2 of IMP.
* Men who were sexually active with partners of childbearing potential and who had not had a verified vasectomy (documented in medical records) that agreed to use condoms with a spermicidal agent and to practice a highly effective form of contraception with their sexual partners born female starting at Visit 0 and continuously until 28 days after receiving the last IMP dose. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only): If 28 days after the participant's first IMP dose had passed before they consent to continue Dose 2, they should have agreed to use condoms with a spermicidal agent and to practice a highly effective form of contraception with their sexual partners born female starting from the time they consent to Dose 2 and continuously until 28 days after receiving Dose 2 of IMP.
* Men who were willing to refrain from sperm donation, starting at Visit 0 and continuously until 28 days after receiving the last IMP dose. Inclusion criteria pertaining to Dose 2 (Cohorts 1-4 only): If 28 days after the participant's first IMP dose had passed before they consent to continue Dose 2, they should have agreed to refrain from sperm donation, starting from the time they consent to Dose 2 and continuously until 28 days after receiving Dose 2 of IMP.

Inclusion Criteria (Dose 2 groups, Cohorts 1-4 only):

Participants were eligible to receive Dose 2 if all of the following criteria (in addition to inclusion criteria above) apply:

* Had given informed consent by signing and dating the ICF reflecting the respective protocol version before administration of Dose 2.
* Had enrolled in a dose cohort and received Dose 1 of BNT162b4 + BNT162b2 Bivalent (original/Omicron BA.4/BA.5) in this trial.
* Were healthy in the opinion of the investigator based on a brief (symptom-directed) physical examination.

Exclusion Criteria (applicable to all dose groups unless specified otherwise):

* Breastfeeding or intending to become pregnant starting with Visit 0 until 28 days after receiving the last dose of trial IMP or intending to father children starting with Visit 0 until 28 days after receiving the last trial IMP dose.
* History of any severe adverse reactions to vaccines or to vaccine components and including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a participant who had an anaphylactic adverse reaction to pertussis vaccine as a child).
* Current or history of the following medical conditions:

  1. Uncontrolled or moderate or severe respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease); symptoms of asthma severity as defined in the most recent US National Heart, Lung, and Blood Institute asthma management guidelines.
  2. Diabetes mellitus type 1 or type 2, or new onset of Diabetes mellitus type 1 or 2 from the administration of Dose 1, including cases controlled with diet alone (Not excluded: history of isolated gestational diabetes).
  3. Hypertension:

     * If a person had been found to have elevated blood pressure or hypertension during screening or previously, excluded for blood pressure that is not well controlled. Well controlled blood pressure was defined as consistently <=140 mm Hg systolic and <= 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤150 mm Hg systolic and ≤90 mm Hg diastolic at Visit 0.
     * If a person did not have a history of elevated blood pressure or hypertension previously or during screening, also excluded for systolic blood pressure ≥150 mm Hg at Visit 0 or diastolic blood pressure ≥100 mm Hg at Visit 0. Exclusion pertaining to Dose 2 (all cohorts): Participants who had new onset of worsening hypertension since enrollment, that, in the opinion of the investigator would constitute an increased risk to the individual's participation in Dose 2 would not receive Dose 2.
  4. Any current or history of cardiovascular diseases such as myocarditis, pericarditis, myocardial infarction, symptomatic congestive heart failure, cardiomyopathy or clinically significant arrhythmias. Exclusion pertaining to Dose 2 (all cohorts): Participants who had new onset of cardiovascular disease since enrollment, that, in the opinion of the investigator would constitute an increased risk to the individual's participation in Dose 2 would not receive Dose 2.
  5. A diagnosed bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions). Exclusion pertaining to Dose 2 (all cohorts): Participants who had new onset of a bleeding disorder since enrollment, that, in the opinion of the investigator, would constitute an increased risk to the individual's participation in Dose 2 would not receive Dose 2.
  6. Seizure disorders: History of seizure(s) within the past 3 years. Also excluded if participant had used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
  7. Screening 12-lead ECG that was consistent with probable or possible myocarditis or pericarditis, or demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of the trial results. Exclusion pertaining to Dose 2 (all cohorts): Only symptomatic participants or whose clinical picture, in the opinion of the investigator, warrant ECG will have a repeat 12-lead ECG prior to Dose 2.

     * Note: ECG changes including but not limited to: paroxysmal or sustained atrial or ventricular arrhythmias, atrioventricular block (grade 2-3) or bundle branch block, diffuse ST-segment elevation or PR-segment inversion, QTcF interval (QT interval corrected by the Fridericia formula) >450 ms in men and >460 ms in women, changes supporting myocardial infarction and/or myocardial ischemia. Exclusion pertaining to Dose 2 (all cohorts): Subjects who had a repeat ECG prior to Dose 2 and had a change or new onset that, in the opinion of the investigator, will not receive Dose 2.
* Current or history of major psychiatric illness, including but not limited to bipolar disorder, major depressive disorder, schizophrenia, autism, and attention deficit-hyperactivity disorder that could interfere with participation and follow-up as required by the trial protocol. Exclusion pertaining to Dose 2 (Cohorts 1-4): Participants who had a change or new onset psychiatric illness.
* Current or history of the following diseases associated with immune dysregulation:

  * Primary immunodeficiencies.
  * History of solid organ or bone marrow transplantation.
  * Asplenia: any condition resulting in the absence of a functional spleen.
  * Currently existing or history of autoimmune disease including and not limited to thyroid autoimmune disease, multiple sclerosis, or psoriasis. Exclusion pertaining to Dose 2 (Cohorts 1-4): Participants who had a change or new onset immunodeficiency.
* Received any non-trial IMP within 28 days before Visit 0 or Visit 7 (Cohorts 1-4) and (Cohort 5) within 28 days before Dose 1 and Dose 2 (except seasonal influenza vaccine, which should be given at least 14 days before or after any administration of IMP).
* Received or planned treatment throughout the entire trial with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for >=14 days at a dose of >=20 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout this trial. Inhaled/nebulized (except high doses as per exclusion criteria above), intraarticular, intrabursal, or topical (skin or eyes) corticosteroids were permitted.
* Blood/plasma products and/or immunoglobulin containing therapy (including monoclonal antibodies) received:

  * Cohorts 1-4: within 120 days before Visit 1 or Visit 7 or administration was planned starting at Visit 0 or prior to Visit 7 until 120 days after the last IMP administration in this trial.
  * Cohort 5: within 120 days before dosing and prior to Dose 2 or administration is planned starting at Visit 0 or prior to Dose 2 until 90 days after the last IMP administration in this trial.
  * Exclusion pertaining to Dose 2 (Cohorts 1-4): if 28 days after the participant's last IMP dose had passed before they consent to continue Dose 2, blood/plasma products and/or immunoglobulin containing therapy (including monoclonal antibodies) received within 120 days before Dose 2 of IMP (Visit 7) continuously until 120 days after receiving Dose 2 of IMP.
* Received allergy treatment with antigen injections within 28 days before Visit 1 or Visit 7 (Cohorts 1-4) and within 28 days before dosing (Cohort 5) or where allergy treatment with antigen injections were scheduled within 14 days after any visit with IMP administration in this trial.
* Participants with a history of SARS-CoV-2 infection (symptomatic or asymptomatic) <60 days prior to randomization.
* Have received any non-RNA or unauthorized COVID-19 vaccine, aside from Dose 1 of the current trial.
* Any existing condition which may affect IMP administration and/or assessment of local reactions assessment at the injection site, e.g., tattoos, severe scars, etc.
* Were vulnerable individuals as per International Council for Harmonisation (ICH) E6 definition, i.e., are individuals whose willingness to participate in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
* Any screening hematology and/or blood chemistry laboratory value that meets the definition of a Grade >=1 abnormality at Visit 0, or an abnormal C-reactive protein (identified by any method) or troponin I value.

  * Note: Participants with any stable Grade 1 abnormalities (according to the toxicity grading scale) may be considered eligible at the discretion of the investigator. Gilberts disease, in and of itself, is not considered exclusionary. Exclusion pertaining to Dose 2: Only symptomatic participants or whose clinical picture, in the opinion of the investigator, warrant laboratory investigation, would have a repeat lab(s) prior to Dose 2.
* History of alcohol abuse or drug addiction within 1 year before Visit 0, or a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their wellbeing if they participate as participants in the trial, or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (17):
- United States (17):
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Hoag Hospital, Newport Beach, California
  - California Research Foundation, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Cenexel RCA (Research Centers of America), Hollywood, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - Great Lakes Clinical Trials LLC - Andersonville, Chicago, Illinois
  - Johnson County Clin-Trials, Inc. (JCCT), Lenexa, Kansas
  - University of Kentucky Center for Clinical and Translational Science (outpatient clinic), Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC (Kansas), Kansas City, Missouri
  - Finger Lakes Clinical Research, Rochester, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Trials of Texas, LLC / Flourish Research, San Antonio, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arieta CM, Xie YJ, Rothenberg DA, Diao H, Harjanto D, Meda S, Marquart K, Koenitzer B, Sciuto TE, Lobo A, Zuiani A, Krumm SA, Cadima Couto CI, Hein S, Heinen AP, Ziegenhals T, Liu-Lupo Y, Vogel AB, Srouji JR, Fesser S, Thanki K, Walzer K, Addona TA, Tureci O, Sahin U, Gaynor RB, Poran A. The T-cell-directed vaccine BNT162b4 encoding conserved non-spike antigens protects animals from severe SARS-CoV-2 infection. Cell. 2023 May 25;186(11):2392-2409.e21. doi: 10.1016/j.cell.2023.04.007. Epub 2023 Apr 13. PMID 37164012
- [Derived] Wang CY, Peng WJ, Kuo BS, Ho YH, Wang MS, Yang YT, Chang PY, Shen YH, Hwang KP. Toward a pan-SARS-CoV-2 vaccine targeting conserved epitopes on spike and non-spike proteins for potent, broad and durable immune responses. PLoS Pathog. 2023 Apr 20;19(4):e1010870. doi: 10.1371/journal.ppat.1010870. eCollection 2023 Apr. PMID 37079651

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years): Participants aged 18-55 years received an intramuscular injection of BNT162b2 Bivalent 30 micrograms (mcg) along with BNT162b4 5 mcg at Day 1.
- Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years): Participants aged greater than (>) 55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 15 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 15 mcg again as Dose 2 at 6 to 7 months after Dose 1.
- Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years): Participants aged > 55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 30 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 30 mcg again as Dose 2 at 6 to 7 months after Dose 1.
Period: Overall Study
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Started | 46 | 45 | 45 | 45 | 46 | 45 | 22 | 59 | 30
Safety Set- Post Dose 1 (Two participants randomized in Cohort 3b received BNT162b2 Bivalent + 5 mcg BNT162b4 treatment in Cohort 1 and were analyzed in Cohort 1 for the safety analysis.) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Safety Set- Post Dose 2 (Cohort 1, Comparator Cohorts A and B did not receive Dose 2 of the study drugs.) | 0 | 30 | 30 | 31 | 37 | 34 | 19 | 0 | 0
Dose 1 (At Day 1) | 46 | 44 | 44 | 45 | 46 | 45 | 21 | 59 | 29
Dose 2 (At 6 Months for Cohorts 1, 2, 3a, 3b,4a, 4b and Comparator Cohorts;at 2 Months for Cohort 5) | 0 | 30 | 30 | 31 | 37 | 34 | 19 | 0 | 0
Completed | 46 | 44 | 44 | 45 | 46 | 45 | 19 | 59 | 29
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Randomized but not dosed | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years) | Total
Number analyzed (Participants) | 46 | 45 | 45 | 45 | 46 | 45 | 22 | 59 | 30 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (10.02) | 40.2 (10.67) | 40.6 (9.67) | 67.3 (5.72) | 40.9 (10.57) | 67.1 (7.14) | 37.9 (11.78) | 38.9 (10.84) | 67.5 (6.57) | 48.8 (15.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 27 | 25 | 24 | 27 | 11 | 31 | 20 | 224
  Male | 16 | 16 | 18 | 20 | 22 | 18 | 11 | 28 | 10 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 16 | 18 | 11 | 14 | 11 | 13 | 22 | 6 | 131
  Not Hispanic or Latino | 26 | 29 | 27 | 34 | 32 | 34 | 9 | 36 | 24 | 251
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 1 | 2 | 0 | 1 | 3 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 3 | 4 | 2 | 4 | 1 | 1 | 3 | 3 | 25
  White | 41 | 37 | 40 | 41 | 39 | 44 | 20 | 50 | 26 | 338
  More than one race | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Reactions- Post Dose 1
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) and pre-listed (that is, solicited) in the e-diary. Solicited local reactions included: pain, erythema/redness, and induration/swelling.
Time Frame: Up to 7 days post-dose1
Population: Analysis was performed on safety set that included all participants who received at least one dose of investigational medicinal product (IMP). Here, overall number of participants analyzed signifies participants with available data for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 42 | 45 | 45 | 21 | 59 | 29
Participants
  Pain | 30 | 30 | 29 | 30 | 41 | 33 | 13 | 35 | 16
  Erythema/Redness | 7 | 3 | 5 | 4 | 2 | 2 | 0 | 4 | 3
  Induration/Swelling | 5 | 5 | 5 | 4 | 2 | 0 | 1 | 3 | 2

2. Primary Outcome: Number of Participants With Solicited Local Reactions- Post Dose 2
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) and pre-listed (that is, solicited) in the e-diary. Solicited local reactions included: pain, erythema/redness, and induration/swelling. Data for this outcome measure was not collected and analyzed for Cohort 1, and Comparator Cohorts A and B, as these Cohorts did not receive Dose 2 of the study drugs.
Time Frame: Up to 7 days post-dose 2
Population: Analysis was performed on dose 2 safety set, that is, all participants who received two doses of IMP. Here, overall number of participants analyzed signifies participants with available data for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 29 | 29 | 31 | 37 | 34 | 19
Participants
  Pain | 23 | 18 | 23 | 29 | 24 | 11
  Erythema/Redness | 2 | 2 | 4 | 3 | 0 | 0
  Induration/Swelling | 2 | 1 | 2 | 3 | 0 | 1

3. Primary Outcome: Number of Participants With Solicited Systemic Events- Post Dose 1
Description: A solicited reaction was defined as an adverse reaction observed and reported under the conditions (symptom and onset) pre-listed (i.e., solicited) in the e-diary. Solicited systemic reactions included: vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, and fever.
Time Frame: Up to 7 days post-dose 1
Population: Analysis was performed on safety set that included all participants who received at least one dose of IMP. Here, overall number of participants analyzed signifies participants with available data for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 42 | 46 | 45 | 21 | 59 | 29
Participants
  Vomiting | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
  Diarrhea | 7 | 3 | 3 | 5 | 2 | 3 | 0 | 3 | 3
  Headache | 16 | 13 | 16 | 13 | 21 | 12 | 3 | 15 | 8
  Fatigue | 24 | 16 | 22 | 21 | 27 | 18 | 5 | 21 | 8
  Myalgia | 21 | 20 | 20 | 15 | 27 | 13 | 8 | 19 | 4
  Arthralgia | 10 | 9 | 6 | 8 | 7 | 6 | 2 | 6 | 0
  Chills | 10 | 11 | 8 | 9 | 12 | 8 | 0 | 8 | 5
  Fever | 3 | 1 | 1 | 4 | 5 | 2 | 0 | 3 | 1

4. Primary Outcome: Number of Participants With Solicited Systemic Events- Post Dose 2
Description: as for outcome 3
Time Frame: Up to 7 days post-dose 2
Population: Analysis was performed on dose 2 safety set. Here, overall number of participants analyzed signifies participants with available data for the analysis. Data for this outcome measure was not collected and analyzed for Cohort 1, and Comparator Cohorts A and B as these Cohorts did not receive Dose 2 of the study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 29 | 29 | 31 | 37 | 34 | 19
Participants
  Vomiting | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea | 1 | 4 | 2 | 3 | 0 | 2
  Headache | 9 | 10 | 10 | 16 | 5 | 3
  Fatigue | 12 | 12 | 16 | 19 | 14 | 8
  Myalgia | 13 | 14 | 9 | 20 | 12 | 5
  Arthralgia | 7 | 6 | 3 | 7 | 7 | 4
  Chills | 7 | 2 | 5 | 14 | 4 | 2
  Fever | 1 | 0 | 1 | 2 | 0 | 1

5. Primary Outcome: Number of Participants With Adverse Events (AEs)-Post Dose 1
Description: An AE was defined as any untoward medical occurrence in a participant administered with a pharmaceutical product, and which did not necessarily have a causal relationship with this treatment.
Time Frame: Up to 28 days post-dose 1
Population: Analysis was performed on safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Participants | 11 | 4 | 8 | 6 | 8 | 5 | 1 | 13 | 5

6. Primary Outcome: Number of Participants With Adverse Events (AEs)-Post Dose 2
Description: as for outcome 5
Time Frame: Up to 28 days post-dose 2
Population: Analysis was performed on dose 2 safety set. Data for this outcome measure was not collected and analyzed for Cohort 1, and Comparator Cohorts A and B as these Cohorts did not receive Dose 2 of the study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants | 3 | 9 | 3 | 5 | 2 | 2

7. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)-Post Dose 1
Description: An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death and was life-threatening. It also included any event requiring hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, caused a congenital anomaly or birth defect, or any other event determined as SAE as per medical or scientific judgment.
Time Frame: Up to 6 to 7 months post-dose 1 for Cohorts 1 to 4 and Comparator Cohorts; and up to 2 months post-dose 1 for Cohort 5
Population: Analysis was performed on safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Participants | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)-Post Dose 2
Description: as for outcome 7
Time Frame: Up to 6 to 7 months post-dose 2 for Cohorts 2 to 4; and up to 3 months post-dose 2 for Cohort 5
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants | 1 | 0 | 1 | 1 | 1 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Hematological Parameters-Post Dose 1
Description: Participants with hematological abnormalities for basophils, eosinophils, erythrocytes, hematocrit, hemoglobin, leukocytes, lymphocytes, monocytes, neutrophils and platelets were analyzed and only clinically significant abnormal data was reported in the outcome measure.
Time Frame: At Day 3 post-Dose 1; at Day 7 post-dose 1
Population: Analysis was performed on safety set. Here, number analyzed signifies participants with available data for each specified category and "0" in the number analyzed field signifies that no participants were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Participants
  Basophils- Day 3 post dose-1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Basophils- Day 3 post dose-1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Basophil-Day 7 post dose-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Eosinophils- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Eosinophils- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Erythrocytes- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Erythrocytes- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Erythrocytes- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Hematocrit- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Hematocrit- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Hemoglobin- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Hemoglobin- Day 7 post-dose 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Leukocytes- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Leukocytes- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Leukocytes- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Lymphocytes- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Lymphocytes- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Monocytes- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Monocytes- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Neutrophils- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Neutrophils- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Platelets- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Platelets- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Hematological Parameters-Post Dose 2
Description: as for outcome 9
Time Frame: At Day 7 post-dose 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants
  Basophils-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Day 7 post dose-2 | 0 | 0 | 0 | 1 | 0 | 0
  Hematocrit-Day 7 post dose-2 | 0 | 0 | 0 | 1 | 0 | 0
  Hemoglobin-Day 7 post dose-2 | 0 | 3 | 0 | 1 | 0 | 0
  Leukocytes-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets-Day 7 post dose-2 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Clinical Chemistry-Post Dose 1
Description: Participants with laboratory abnormalities (clinical chemistry) for alanine aminotransferase, albumin, alkaline phosphatase, amylase, aspartate aminotransferase, C-reactive protein, creatinine, direct bilirubin, gamma glutamyl transferase, glucose, high sensitivity C reactive protein, indirect bilirubin, lipase, total bilirubin, troponin I type 3 and urea nitrogen were analyzed and only abnormal clinically significant data was reported in the outcome measure.
Time Frame: At Day 3 post-Dose 1; at Day 7 post-dose 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Participants
  Alanine Aminotransferase- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Alanine Aminotransferase- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Alanine Aminotransferase- Day 7 post-dose 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
  Albumin- Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Albumin- Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Albumin- Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase-Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Alkaline Phosphatase-Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Alkaline Phosphatase-Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Amylase- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Amylase- Day 7 post dose 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Aspartate Aminotransferase- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Aspartate Aminotransferase- Day 7 post dose 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  C Reactive Protein- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  C Reactive Protein- Day 3 post dose 1 | 0 | 1 | 0 |  | 0 |  |  | 0 |
  C Reactive Protein- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Creatinine- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Creatinine- Day 7 post dose 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Direct Bilirubin- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Direct Bilirubin- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Gamma Glutamyl Transferase- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Gamma Glutamyl Transferase- Day 7 post dose 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Glucose- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Glucose- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Glucose- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  High Sensitivity C Reactive Protein- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  High Sensitivity C Reactive Protein- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  High Sensitivity C Reactive Protein- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Indirect Bilirubin- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Indirect Bilirubin- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Lipase- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Lipase- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Total Bilirubin- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Total Bilirubin- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Total Bilirubin- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I Type 3- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Troponin I Type 3- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Troponin I Type 3- Day 7 post dose 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen- Day 3 post dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Urea Nitrogen- Day 3 post dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Urea Nitrogen- Day 7 post dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Clinical Chemistry-Post Dose 2
Description: Participants with laboratory abnormalities (clinical chemistry) for alanine aminotransferase, albumin, alkaline phosphatase, amylase, aspartate aminotransferase, C-reactive protein, creatinine, direct bilirubin, gamma glutamyl transferase, glucose, high sensitivity C reactive protein, indirect bilirubin, lipase, total bilirubin, troponin I type 3 and urea nitrogen were analyzed and only clinically significant abnormal data was reported in the outcome measure.
Time Frame: At Day 7 post-dose 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants
  Alanine Aminotransferase-Day 7 post-dose 2 | 0 | 0 | 0 | 1 | 0 | 0
  Albumin-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase-Day 7 post-dose 2 | 0 | 0 | 0 | 1 | 0 | 0
  C Reactive Protein-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase-Day 7 post-dose 2 | 0 | 0 | 0 | 1 | 0 | 0
  Glucose-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  High Sensitivity C Reactive Protein-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I Type 3-Day 7 post-dose 2 | 0 | 1 | 0 | 0 | 0 | 0
  Urea Nitrogen-Day 7 post-dose 2 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Clinically Significant New Electrocardiogram (ECG) Abnormalities -Post Dose 1
Description: Participants with only clinically significant new ECG abnormalities were reported in the outcome measure.
Time Frame: At Day 3 post-Dose 1; at Day 7 post-dose 1
Population: Analysis was performed on safety set. Here, overall number of participants analyzed signifies participants with available data for the analysis and number analyzed signifies participants with available data for each specified category and "0" in the number analyzed field signifies that no participants were available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 47 | 43 | 43 | 42 | 46 | 44 | 21 | 59 | 29
Participants
  Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 8 | 59 | 0
  Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  | 0 | 0 |
  Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Clinically Significant New ECG Abnormalities -Post Dose 2
Description: Participants with only clinically significant new ECG abnormalities were reported in the outcome measure.
Time Frame: At Day 7 post-dose 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years): Participants aged 18-55 years received an intramuscular injection of BNT162b2 Bivalent 30 mcg along with BNT162b4 10 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Bivalent 30 mcg along with BNT162b4 10 mcg again as Dose 2, 6 to 7 months after Dose 1.
- Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years): Participants aged 18-55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 15 mcg at Day 1, Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 15 mcg again as Dose 2, 6 to 7 months after Dose 1.
- Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years): Participants aged >55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 15 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 15 mcg again as Dose 2, 6 to 7 months after Dose 1.
- Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years): Participants aged 18-55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 30 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 30 mcg again as Dose 2, 6 to 7 months after Dose 1.
- Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years): Participants aged >55 years received a dose of BNT162b2 Bivalent 30 mcg (Omicron BA.4/BA.5) along with BNT162b4 30 mcg at Day 1. Participants who consented to receive a second dose of the study drugs received BNT162b2 Monovalent (OMI XBB.1.5) 30 mcg along with BNT162b4 30 mcg again as Dose 2, 6 to 7 months after Dose 1.
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Shift of Laboratory Parameters (Hematology) From Baseline Grade 0 to Worst Grade >=3: Post-dose 1
Description: The intensity of AEs and laboratory parameters was graded by the investigator. Grades were defined as: Grade 1 - Mild; does not interfere with the trial participant's usual function; Grade 2 - Moderate; interferes to some extent with the trial participant's usual function; Grade 3 - Severe; interferes significantly with the trial participant's usual function and Grade 4 - Potentially life-threatening; life-threatening consequences, urgent intervention required. Participants with shift change from Baseline Grade 0 to Worst Grade >=3 were reported in the outcome measure.
Time Frame: At Day 3 post-dose 1; at Day 7 post-dose 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Participants
  Eosinophils-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 5 | 0 | 6 | 0 | 0 | 8 | 0
  Eosinophils-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Eosinophils-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1: number analyzed (Participants) | 45 | 42 | 43 | 42 | 44 | 43 | 20 | 57 | 29
  Eosinophils-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 0
  Hemoglobin-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 |  | 0 |  | 0 |  |  | 0 |
  Hemoglobin-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1: number analyzed (Participants) | 10 | 11 | 15 | 5 | 5 | 5 | 3 | 12 | 3
  Hemoglobin-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes-White blood cell decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Leukocytes-White blood cell decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Leukocytes-White blood cell decreased-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes-White blood cell increased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Leukocytes-White blood cell increased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Leukocytes-White blood cell increased-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes count decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Lymphocytes count decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Lymphocytes count decreased-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Neutrophil count decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Neutrophil count decreased-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Platelet count decreased-Baseline Grade 0 to Grade >=3: Day 3 post-Dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Platelet count decreased-Baseline Grade 0 to Grade >=3: Day 7 post-Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Number of Participants With Shift of Laboratory Parameters (Hematology) From Baseline Grade 0 to Worst Grade >=3: Post Dose 2
Description: as for outcome 15
Time Frame: At Day 7 post-dose 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants
  Eosinophils-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Baseline Grade 0 to Grade >=3 | 0 | 1 | 1 | 2 | 2 | 0
  Leukocytes-White blood cell decreased-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes-White blood cell increased-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes count decreased-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Shift of Laboratory Parameters (Clinical Chemistry) From Baseline Grade 0 to Worst Grade >=3: Post Dose 1
Description: as for outcome 15
Time Frame: At Day 3 post-dose 1; at Day 7 post-dose 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 48 | 44 | 44 | 43 | 46 | 45 | 21 | 59 | 29
Participants
  Alanine Aminotransferase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Alanine Aminotransferase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Alanine Aminotransferase: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Albumin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Albumin: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Alkaline Phosphatase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Alkaline Phosphatase: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Amylase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Amylase: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Aspartate Aminotransferase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Aspartate Aminotransferase: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Creatinine: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Creatinine: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Direct Bilirubin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Direct Bilirubin: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Glucose: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Glucose: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Indirect Bilirubin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Indirect Bilirubin: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Lipase: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Lipase: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Total Bilirubin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Total Bilirubin: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Total Bilirubin: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1: number analyzed (Participants) | 6 | 6 | 6 | 0 | 6 | 0 | 0 | 8 | 0
  Urea Nitrogen: Baseline Grade 0 to Grade >=3 Day 3 post-dose 1 | 0 | 0 | 0 |  | 0 |  |  | 0 |
  Urea Nitrogen: Baseline Grade 0 to Grade >=3 Day 7 post-dose 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Shift of Laboratory Parameters (Clinical Chemistry) From Baseline Grade 0 to Worst Grade >=3: Post-dose 2
Description: as for outcome 15
Time Frame: At Day 7 post-dose 2
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 30 | 30 | 31 | 37 | 34 | 19
Participants
  Alanine aminotransferase-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Serum amylase-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase-Baseline Grade 0 to Grade >=3 | 0 | 0 | 1 | 0 | 0 | 0
  Total Bilirubin-Baseline Grade 0 to Grade >=3 | 0 | 0 | 0 | 0 | 0 | 0
  Blood urea nitrogen-Baseline Grade 0 to Grade >=3 | 0 | 0 | 1 | 0 | 0 | 0

19. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 Neutralizing Antibody Ancestral Strain-Post Dose 1
Description: GMTs for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) neutralizing antibody ancestral strain were measured by valid assay method. Data for this outcome measure was not planned to be collected and analyzed for Cohort 5.
Time Frame: At Pre-dose and Day 28 post dose-1
Population: Analysis was performed on Immunogenicity per protocol set that is all participants who received the planned dose of the IMP on Day 1 and who have at least one valid immunogenicity assessment within an appropriate window and have no major protocol deviations that can confound immunogenicity data. Here, overall number of participants analyzed signifies participants with available data for the analysis and number analyzed signifies participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 44 | 41 | 44 | 42 | 46 | 44 | 58 | 29
titers
  Pre-dose | 3310.0 [2404.0 to 4557.4] | 4561.4 [3036.1 to 6853.2] | 3031.5 [1962.7 to 4682.3] | 6245.1 [4446.8 to 8770.5] | 3052.9 [2115.7 to 4405.3] | 2267.0 [1599.6 to 3212.8] | 3579.9 [2447.0 to 5237.3] | 4034.9 [2321.9 to 7011.7]
  28 days post-dose 1: number analyzed (Participants) | 40 | 39 | 42 | 40 | 39 | 41 | 56 | 29
  28 days post-dose 1 | 12666.7 [9744.2 to 16465.6] | 13017.3 [9639.5 to 17578.7] | 9571.7 [7120.1 to 12867.4] | 14553.1 [11441.6 to 18510.9] | 10326.7 [7827.3 to 13624.4] | 10126.2 [7730.8 to 13263.9] | 12767.2 [9848.9 to 16550.1] | 14628.7 [10394.8 to 20587.0]

20. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 Neutralizing Antibody Ancestral Strain-Post Dose 2
Description: GMTs for SARS-CoV-2 neutralizing antibody ancestral strain were measured by valid assay method. Data for this outcome measure was not planned to be collected and analyzed for Cohort 5.
Time Frame: At Pre-dose 2 and Day 28 post-dose 2
Population: Analysis was performed on Immunogenicity per protocol set. Here, overall number of participants analyzed signifies participants with available data for the analysis and number analyzed signifies participants with available data for each specified category and "0" in the number analyzed field signifies that no participants were available for the analysis at the specified time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 38 | 33 | 39 | 37 | 36 | 30 | 55 | 27
titers
  Pre-Dose-2 | 5940.9 [4413.3 to 7997.2] | 5717.3 [3725.5 to 8774.0] | 3559.2 [2495.8 to 5075.6] | 5751.4 [4322.6 to 7652.5] | 3862.0 [2713.4 to 5496.7] | 3551.6 [2392.2 to 5272.9] | 5238.7 [3869.6 to 7092.2] | 5490.6 [3394.2 to 8881.9]
  28 days post-dose 2: number analyzed (Participants) | 0 | 25 | 25 | 28 | 26 | 22 | 0 | 0
  28 days post-dose 2 |  | 10032.4 [6551.6 to 15362.6] | 7329.5 [4942.9 to 10868.6] | 12884.0 [9244.3 to 17956.7] | 7782.0 [4992.9 to 12129.2] | 6294.6 [3683.9 to 10755.4] |  |

21. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 Neutralizing Antibody Omicron Strains (SARS-CoV-2 Omicron BA.4/BA.5)- Post Dose 1
Description: GMTs for SARS-CoV-2 Omicron BA.4/BA.5 strain were measured by valid assay method.
Time Frame: At Pre-dose and Day 28 post-dose 1
Population: Analysis was performed on immunogenicity per protocol set. Here, number analyzed signifies participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Cohort 5.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 44 | 41 | 44 | 42 | 46 | 44 | 58 | 29
titers
  Pre-dose | 881.7 [553.4 to 1404.5] | 1475.9 [893.5 to 2438.1] | 1125.3 [692.1 to 1829.5] | 1948.8 [1250.3 to 3037.6] | 1067.2 [739.1 to 1541.1] | 625.2 [406.8 to 961.0] | 1485.1 [993.4 to 2220.1] | 1213.0 [665.0 to 2212.8]
  28 days post-dose 1: number analyzed (Participants) | 40 | 39 | 42 | 40 | 39 | 41 | 56 | 29
  28 days post-dose 1 | 5540.9 [3878.4 to 7916.1] | 6801.2 [5000.7 to 9249.9] | 4690.6 [3313.1 to 6640.9] | 6303.1 [4775.2 to 8319.8] | 5913.9 [4330.8 to 8075.8] | 3907.0 [2802.3 to 5447.3] | 6323.4 [4390.6 to 9107.0] | 6552.0 [3927.7 to 10929.8]

22. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 Neutralizing Antibody Omicron Strains (SARS-CoV-2 Omicron BA.4/BA.5)- Post Dose 2
Description: GMTs for SARS-CoV-2 Omicron BA.4/BA.5 strain were measured by valid assay method. Data for this outcome measure was not planned to be collected and analyzed for Cohort 5.
Time Frame: At Pre-dose 2 and Day 28 post-dose 2
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 38 | 33 | 39 | 37 | 36 | 30 | 55 | 27
titers
  Pre-dose-2 | 2597.0 [1733.5 to 3890.5] | 2502.1 [1563.8 to 4003.6] | 1750.6 [1223.9 to 2504.1] | 2089.7 [1422.2 to 3070.4] | 2179.6 [1583.2 to 3000.7] | 1663.4 [1057.0 to 2617.8] | 2649.8 [1906.0 to 3683.8] | 2610.0 [1427.1 to 4773.3]
  28 days post-dose 2: number analyzed (Participants) | 0 | 25 | 0 | 0 | 0 | 0 | 0 | 0
  28 days post-dose 2 |  | 6506.3 [4270.1 to 9913.7] |  |  |  |  |  |

23. Secondary Outcome: Geometric Mean Titers (GMTs) for SARS-CoV-2 Neutralizing Antibody Omicron Strains (SARS-CoV-2 Omicron XBB1.5)- Post Dose 2
Description: GMTs for SARS-CoV-2 Omicron XBB1.5 strain were measured by valid assay method.
Time Frame: At Pre-dose 2 and Day 28 post-dose 2
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number of participants analyzed signifies participants with available data for the analysis and number analyzed signifies participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for Cohorts 1, 2, 5 and Comparator Cohorts A and B.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 39 | 37 | 37 | 31
titers
  Pre-dose-2 | 353.3 [227.1 to 549.6] | 356.8 [219.8 to 579.0] | 608.2 [413.8 to 894.0] | 335.2 [199.1 to 564.4]
  28 days post-dose 2: number analyzed (Participants) | 25 | 28 | 26 | 22
  28 days post-dose 2 | 2493.1 [1572.4 to 3953.0] | 3325.2 [2110.1 to 5239.8] | 3042.7 [1850.6 to 5002.5] | 1935.9 [1061.7 to 3530.1]

24. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 Ancestral Strain-Post Dose 1
Description: GMFRs are defined as ratios of the results after vaccination (that is 28 days post-dose 1) to the results before vaccination (that is pre-dose 1).
Time Frame: From pre-dose 1 to 28 days post-dose 1
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number analyzed signifies participants with available data for the analysis. Data for this outcome measure was not planned to be collected and analyzed for Cohorts 5.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 40 | 39 | 42 | 40 | 39 | 41 | 56 | 29
ratio | 3.4 [2.7 to 4.4] | 2.9 [2.1 to 4.0] | 3.3 [2.4 to 4.6] | 2.3 [1.8 to 3.1] | 3.4 [2.6 to 4.5] | 4.2 [3.2 to 5.5] | 3.7 [2.8 to 4.9] | 3.6 [2.3 to 5.7]

25. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 Ancestral Strain-Post Dose 2
Description: GMFRs are defined as ratios of the results after vaccination (that is 28 days post-dose 2) to the results before vaccination (that is pre-dose 2). Data for this outcome measure was not planned to be collected and analyzed for Cohorts 1, 5 and Comparator Cohorts A and B.
Time Frame: From pre-dose 2 to 28 days post-dose 2
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number analyzed signifies participants with available data for the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 25 | 25 | 28 | 26 | 22
ratio | 2.2 [1.4 to 3.6] | 2.0 [1.2 to 3.5] | 2.1 [1.4 to 3.0] | 2.6 [1.8 to 3.6] | 2.8 [1.7 to 4.7]

26. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 Omicron Strain (OMI BA.4/BA.5)-Post Dose 1
Description: as for outcome 24
Time Frame: From pre-dose 1 to 28 days post-dose 1
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number analyzed signifies participants with available data for the analysis. Data for this outcome measure was not planned to be collected and analyzed for Cohort 5.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 40 | 39 | 42 | 40 | 39 | 41 | 56 | 29
ratio | 5.4 [3.6 to 8.1] | 4.5 [3.0 to 6.8] | 4.4 [3.0 to 6.5] | 3.1 [2.2 to 4.4] | 5.8 [4.3 to 7.8] | 5.9 [4.2 to 8.2] | 4.3 [3.2 to 5.7] | 5.4 [3.4 to 8.7]

27. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 Omicron Strain (OMI BA.4/BA.5)-Post Dose 2
Description: GMFRs are defined as ratios of the results after vaccination (that is 28 days post-dose 2) to the results before vaccination (that is pre-dose 2).
Time Frame: From pre-dose 2 to 28 days post-dose 2
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number analyzed signifies participants with available data for the analysis. Data for this outcome measure was not planned to be collected and analyzed for Cohorts 1, 3a and 3b, 4a and 4b, 5 and Comparator Cohorts A and B.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 25
ratio | 4.4 [2.4 to 8.0]

28. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for SARS-CoV-2 Omicron Strain (Omicron XBB1.5)-Post Dose 2
Description: as for outcome 27
Time Frame: From Pre-dose 2 to Day 28 post-dose 2
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number analyzed signifies participants with available data for the analysis. Data for this outcome measure was not planned to be collected and analyzed for Cohorts 1, 2, 5 and Comparator Cohorts A and B.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 25 | 27 | 26 | 22
ratio | 5.6 [3.7 to 8.5] | 7.8 [5.5 to 11.1] | 4.9 [3.2 to 7.4] | 6.5 [4.2 to 10.2]

29. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Ancestral Strain-Post Dose 1
Description: Seroresponse was defined as achieving >=4-fold rise from baseline (that is, pre-dose).
Time Frame: At Day 28 post-dose 1
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 40 | 39 | 42 | 40 | 39 | 41 | 56 | 29
percentage of participants | 32.5 [18.6 to 49.1] | 30.8 [17.0 to 47.6] | 35.7 [21.6 to 52.0] | 20.0 [9.1 to 35.6] | 38.5 [23.4 to 55.4] | 43.9 [28.5 to 60.3] | 50.0 [36.3 to 63.7] | 41.4 [23.5 to 61.1]

30. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Ancestral Strain-Post Dose 2
Description: Seroresponse was defined as achieving >=4-fold rise from baseline (that is, pre-dose).
Time Frame: At Day 28 post-dose 2
Population: Analysis was performed on immunogenicity per protocol set. Here, overall number analyzed signifies participants with available data for the analysis. Data for this outcome measure was not planned to be collected and analyzed for Cohorts, 1, 5 and Comparator Cohorts A and B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 25 | 25 | 28 | 26 | 22
percentage of participants | 24.0 [9.4 to 45.1] | 16.0 [4.5 to 36.1] | 32.1 [15.9 to 52.4] | 23.1 [9.0 to 43.6] | 27.3 [10.7 to 50.2]

31. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strains (OMI BA.4/BA.5)- Post Dose 1
Description: Seroresponse was defined as achieving >=4-fold rise from baseline (that is, pre-dose).
Time Frame: At Day 28 post-dose 1
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 40 | 39 | 42 | 40 | 39 | 41 | 56 | 29
percentage of participants | 52.5 [36.1 to 68.5] | 46.2 [30.1 to 62.8] | 47.6 [32.0 to 63.6] | 30.0 [16.6 to 46.5] | 59.0 [42.1 to 74.4] | 61.0 [44.5 to 75.8] | 44.6 [31.3 to 58.5] | 55.2 [35.7 to 73.6]

32. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strains (OMI BA.4/BA.5)- Post Dose 2
Description: Seroresponse was defined as achieving >=4-fold rise from baseline (that is, pre-dose).
Time Frame: At Day 28 post-dose 2
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years)
Number analyzed (Participants) | 25
percentage of participants | 44.0 [24.4 to 65.1]

33. Secondary Outcome: Percentage of Participants With Seroresponse to SARS-CoV-2 Omicron Strains (SARS-CoV-2 Omicron XBB1.5)- Post Dose 2
Description: Seroresponse was defined as achieving >=4-fold rise from baseline (that is, pre-dose).
Time Frame: At Day 28 post-dose 2
Population: as for outcome 28
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years)
Number analyzed (Participants) | 44 | 42 | 46 | 44
percentage of participants | 64.0 [42.5 to 82.0] | 77.8 [57.7 to 91.4] | 50.0 [29.9 to 70.1] | 72.7 [49.8 to 89.3]

ADVERSE EVENTS:
Time Frame: AE data was collected from Day 1 up to 28 days post each dose. All SAE data collected throughout the study were reported in AE section and were collected from up to 6 to 7 months post-dose 1 for Cohorts 1 to 4 and Comparator Cohorts; and 6 to 7 months post-dose 2 for Cohorts 2 to 4. For Cohort 5, SAEs: from IMP Dose 1 up to 2 months after Dose 1 and from IMP Dose 2 up to 3 months after Dose 2
Description: Analysis was performed on safety set. Per protocol, solicited local and systemic reactions were not included in the AE analysis unless they continued longer than 7 days post-IMP administration or were a SAE. These reactions are presented in the respective outcome measures. Two participants randomized in Cohort 3b received BNT162b2 Bivalent + BNT162b4 5 mcg treatment in Cohort 1 and were analyzed in Cohort 1 for safety analysis.
Groups:
- Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years: Participants aged 18-55 years received an intramuscular injection of BNT162b2 Bivalent 30 mcg along with BNT162b4 5 mcg at Day 1.
Arm/Group | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/44 | 0/44 | 0/46 | 0/59 | 0/21 | 0/43 | 0/45 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/44 | 1/44 | 1/46 | 1/59 | 0/21 | 2/43 | 1/45 | 0/29
Other Adverse Events (participants affected / at risk) | 3/48 | 1/44 | 1/44 | 6/46 | 1/59 | 0/21 | 4/43 | 10/45 | 1/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years (N=48) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) (N=44) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) (N=44) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) (N=46) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) (N=59) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) (N=21) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) (N=43) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) (N=45) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years) (N=29)
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord herniation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BNT162b2 Bivalent 30 mcg + BNT162b4 5 mcg (Aged 18-55 Years (N=48) | Cohort 2: BNT162b2 Bivalent 30 mcg + BNT162b4 10 mcg (Aged 18-55 Years) (N=44) | Cohort 3a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged 18-55 Years) (N=44) | Cohort 4a: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged 18-55 Years) (N=46) | Comparator A: BNT162b2 Bivalent 30 mcg (Aged 18-55 Years) (N=59) | Cohort 5: BNT162b4 30 mcg (Aged 18-55 Years) (N=21) | Cohort 3b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 15 mcg (Aged >55 Years) (N=43) | Cohort 4b: BNT162b2 Bivalent/Monovalent 30 mcg + BNT162b4 30 mcg (Aged >55 Years) (N=45) | Comparator B: BNT162b2 Bivalent 30 mcg (Aged >55 Years) (N=29)
COVID-19 (Infections and infestations) | 0 | 1 | 1 | 5 | 0 | 0 | 4 | 10 | 1
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 — Also includes solicited systemic reactions that continued longer than 7 days post-IMP administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT05541861/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT05541861/SAP_001.pdf